# Dispatcher-Assisted Cardiopulmonary Resuscitation: A Randomized Controlled Trial of Low-Dose, High-Frequency Simulation-Based Training and the Impact on Real Out-of-Hospital Cardiac Arrest Calls

### **General Information**

Primary Sponsor and Principal Investigator: Freddy Lippert, MD, Associate Professor, Copenhagen Emergency Medical Services, and The Faculty of Health and Medical Sciences, Department of Clinical Medicine, University of Copenhagen, Denmark

Responsible Investigator: Freddy Lippert, MD, Associate Professor

Funding: The study is financed by an unrestricted research grant from the Danish foundation TrygFonden.

#### **Trial registration**

The protocol will be registered on ClinicalTrials.gov prior to enrolment and randomisation of participants. All items from the World Health Organization Trial Registration Data Set will be reported.

#### **Investigators:**

Oscar Rosenkrantz, Copenhagen Emergency Medical Services, and Copenhagen Academy for Medical Education and Simulation, Capital Region of Denmark and University of Copenhagen, Copenhagen, Denmark Kristine Elisabeth Eberhard, Copenhagen Emergency Medical Services, and Copenhagen Academy for Medical Education and Simulation, Capital Region of Denmark and University of Copenhagen, Copenhagen, Denmark Roselil Maria Oelrich, Copenhagen Emergency Medical Services, University of Copenhagen, Copenhagen, Denmark

Anne Lippert, Copenhagen Academy for Medical Education and Simulation, Capital Region of Denmark and University of Copenhagen, Copenhagen, Denmark

Gitte Linderoth, Copenhagen Emergency Medical Services, and Department of Anaesthesia and Intensive Care, Copenhagen University Hospital – Bispebjerg and Frederiksberg Hospital, Copenhagen, Denmark Anders Granholm, Department of Intensive Care 4131, Copenhagen University Hospital – Rigshospitalet, Copenhagen, Denmark

Annette Kjær Ersbøll, National Institute of Public Health, University of Southern Denmark, Copenhagen, Denmark

Fredrik Folke, Copenhagen Emergency Medical Services, and Herlev Gentofte Hospital, Department of Cardiology, and The Faculty of Health and Medical Sciences, Department of Clinical Medicine, University of Copenhagen, Denmark

Participants will be enrolled and randomized in the start of September 2019.

Data collection is planned to start in mid-September 2019 and run for 13 weeks.

## Supplementary assessment points for table 1 – questionnaire content for simulated and real OHCA calls

| | Result (time or |
|---|---|
| Assessment points | yes/no/NA) |
| Address verified? | (yes/no) |
| Patient placed on hard surface? | (yes/no) |
| Callers phone set to speaker mode? | (yes/no) |
| Caller guiding in rescue breaths when caller has not received BLS training? | (yes/no) |
| Straight arms addressed? | (yes/no) |
| Hand placement addressed? | (yes/no) |
| Callers placement next to patient addressed? | (yes/no) |